CLINICAL TRIAL: NCT03535025
Title: Postoperative Quality of Recovery in Patients Receiving Anaesthesia: A Prospective Observational Study
Brief Title: Postoperative Quality of Recovery in Patients Receiving Anaesthesia
Status: Completed | Type: Observational
Sponsor: B.P. Koirala Institute of Health Sciences (Other)
Responsible Party: Principal Investigator, Sachin Koirala, Junior Resident, B.P. Koirala Institute of Health Sciences
Other Study IDs: IRC/1090/017
Record Dates: First submitted 2018-04-15; First posted 2018-05-24 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Elective Surgeries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigator's study is designed to evaluate the recovery of patients receiving anaesthesia for surgeries; in different domains like the physiological, nociceptive, cognitive and emotional to the participants' preoperative state.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 18 years or over who are undergoing surgery with anesthesia

Exclusion Criteria:

* Inability to complete the baseline questionnaire for any reason as assessed by the examiner
* Patient with any current psychiatric disturbance
* Patient undergoing a neuropsychological procedure that may impair their ability to participate in the assessment
* Patients undergoing emergency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients above the age of 18yrs under going elective surgery under anaesthesia
Sampling Method: Non-Probability Sample
Enrollment: 195 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
quality of recovery from anaesthesia | 24 hours post operatively
  include the quality of recovery in each domain over the postoperative follow-up period as compared to the same in preoperative period (baseline value) using the postoperative quality of recovery scale. The different domains include physiological (with subdomains: systolic blood pressure, heart rate, temperature, respiratory rate, oxygen requirement, airway, agitation, consciousness and ability to lift head, each scoring from 1 to 3), nociceptive ( scoring 1to 5, higher score means more pain), emotional (1 to 5), activity of daily living( 1 to 3), cognitive ( with subdomains orientation(1 to 3), number forward and backward(1 to 6), word task and executive memory) and impact on ability to work(1 to 3)

SECONDARY OUTCOMES:
factors delaying recovery | 24 hrs post operatively
  factors associated with delay in recovery from anaesthesia for surgery

CONTACTS AND LOCATIONS:
Locations (1):
- BPKIHS, Dharān, Sunsari, Nepal